CLINICAL TRIAL: NCT03514082
Title: Effect of Conservative Treatment on Pulmonary Functions, Gait Oxygen Consumption Balance and Lower Limb Load Distribution in Adolescents With Idiopathic Scoliosis
Brief Title: Oxygen Consumption in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Yasin YURT, Assistant Professor, Eastern Mediterranean University
Other Study IDs: ETK00-2016-0141
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis: Subjects with AIS who are beginning to the conservative treatment.
  Interventions: Device: Rigid Thermoplastic Spinal Brace

INTERVENTIONS:
Device: Rigid Thermoplastic Spinal Brace — Custom made rigid thermoplastic brace with 23 hours daily wearing time.

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a rotational deformity of the spine that could be seen 2-3% of population. Conservative treatment of AIS with 20-45 degree lateral flexion angle (Cobb) includes brace and therapeutic exercises. Some gait abnormalities were defined like decreased torsional movements of spine, increased muscular work and energy expenditure in AIS. Additionally wearing a brace limits pelvic motions and affects pendulum-like mechanism of gait. Our aim was to investigate gait energy consumption, pulmonary functions, balance and lower extremity loading symmetry in AIS subjects who are getting conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cobb angle between 20-45 degree,
* Prescribed a rigid spinal brace by doctor

Exclusion Criteria:

* Having leg length discrepancy more than 1 centimeter
* Having a lung disease
* Having another orthopedic or neurologic disorder

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subject who come to our outpatient clinic will be assessed for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Gait Oxygen Consumption | Assessment will be done at the end of first month of conservative treatment.
  Oxygen consumption will be assessed with a mobile metabolic analyzer during walking on treadmill with 4 km/h gait speed. Recordings will be taken for 2 minutes after first 2 minutes of walking.

SECONDARY OUTCOMES:
Pulmonary Functions | Assessment will be done at the end of first month of conservative treatment.
  Forced vital capacity (FVC), Forced expiratory volume in one second (FEV1), FEV1/FVC ratio, peak expiratory flow (PEF), forced expiratory flow at 25-75 % of the pulmonary volume (FEF 25-75%) will be assessed with spirometer.
Balance | Assessment will be done at the end of first month of conservative treatment.
  Balance will be assessed with a special equipment that gives deviation that lower values mean better.
Lower extremity loading symmetry | Assessment will be done at the end of first month of conservative treatment.
  Plantar loading symmetry will be assessed with a pedobarograph located in the middle of a six meters walking way. Loading symmetry will be calculated and compared as percentage of total pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Yurt, Asst. Prof., Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No